CLINICAL TRIAL: NCT01678859
Title: Cervical Mucus - the Biochemical and Molecular Properties in Fertile and Subfertile Women
Brief Title: Cervical Mucus - the Biochemical and Molecular Properties in Fertile and Subfertile Women (C-MIS Study)
Acronym: C-MIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Merrion Fertility Clinic (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Sponsor
Other Study IDs: MFC 1
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Infertility
Keywords: infertility; cervical; mucus; sperm; interaction
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cervical mucus serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Infertility affects approximately one in six couples1. In approximately one third of cases, there is no cause found as to why a couple are unable to conceive2. In order for natural pregnancy to occur, sperm must pass through the cervix (neck of the womb) and swim to the woman's Fallopian tubes so that fertilisation of one of the woman's eggs can occur. It is known that mid-cycle mucus at the cervix is essential for sperm to gain access to the uterus and tubes.

There is evidence that the composition of this mucus in women may affect fertility but this area has not been studied well in recent years, partly because fertility treatments such as IVF bypass the cervix.

Research in sheep and cows in UCD has shown interesting differences in the cervical mucus of fertile and infertile animals. It appears that the mucus not only helps sperm to get to the uterus but may also help the sperm to mature and be ready to fertilise an egg. This mucus may also help prevent bacteria and infection reaching the womb.

In conjunction with colleagues in UCD, under the leadership of Professor S Carrington, the investigators would like to investigate some of the properties of human cervical mucus.The investigators propose to do this by taking samples of cervical mucus around the time of ovulation and also approximately one week later in fertile women and sub-fertile women. Then to monitor ovulation with an ultrasound scan (follicle tracking) of the woman's ovaries and urinary ovulation kits and take blood for oestrogen, progesterone, LH and FSH levels.

The investigators wish to determine if there are differences between the mucus of these women and how it may impact on sperm function and on fertility.

DETAILED DESCRIPTION:
This study will investigate functional, biochemical and molecular properties of cervical mucus at various times of the menstrual cycle in fertile and sub-fertile women. The investigators would aim to also investigate the interaction of cervical mucus with sperm and capacitation and to investigate the impact cervical surgery and differing diagnoses of sub-fertility have on cervical mucus.

Study aims:

1. To determine the functional, biochemical and molecular properties of cervical mucus through out the menstrual cycle in fertile women.
2. To determine if there is a difference in these properties of cervical mucus in fertile and sub-fertile women.
3. To determine whether these properties are influenced by the sub-fertility diagnostic group eg unexplained, endometriosis, tubal factor, sperm factor.
4. To examine the interaction between cervical mucus and sperm in women with normal fertility and sub-fertility.
5. To examine the impact of cervical surgery on cervical mucus functional, biochemical and molecular properties and sperm interaction.

ELIGIBILITY:
Inclusion Criteria:

1. Fertile women

   1. Age 18-42 years
   2. Regular ovulatory menstrual cycle
   3. Previous spontaneous pregnancy to term
   4. No history of subfertility
   5. No underlying medical condition or immunosuppression
   6. No history of hormonal medication or pregnancy in past two months
   7. Capable of giving informed consent to participate in study
2. Non fertile women a.Age 18-42 years b.Regular ovulatory menstrual cycle c.Difficulty conceiving for greater than 12 months e.No underlying medical condition or immunosuppression f.No history of hormonal medication in past two months g.Capable of giving informed consent to participate in study

Exclusion Criteria:

1. hormonal medication
2. pregnancy
3. not capable of giving consent
4. age <18 years or > 42 years
5. underlying medical condition

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: gyanecological outpatient department
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The ability of sperm to swim through cervical mucus | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: mary wingfield, MD, FRCOG, Principal Investigator — merrion fertility clinic/National Maternity Hospital
Locations (1):
- Merrion fertility clinic/national maternity hospital, Holles Streetdublin 2, Ireland, Dublin 2, Ireland